CLINICAL TRIAL: NCT06397547
Title: The Impact of Flipped Learning Model on Nursing Students' Thorax and Heart Examination Knowledge and Self-directed Learning Skills: A Randomized Controlled Study
Brief Title: Flipped Learning Model on Nursing Students' Thorax and Heart Examination
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Thorax and Heart Examination
Record Dates: First submitted 2024-04-30; First posted 2024-05-03 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Nursing Students; Nursing Caries; Nurse's Role

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flipped learning (Experimental): The experimental group will receive digital materials (such as explanatory and demonstration videos, Edpuzzle, etc.) prior to the topic. The links to these materials will be sent to the students, who can access them via their mobile phones and watch the explanatory and demonstration videos as many times as they wish.
  Subsequently, the topic "Thorax and Heart Examination" will be presented to the students. They will summarize the information learned from the videos and engage in question-answer sessions and discussions using prepared digital resources to address any points they do not understand. To reinforce the practices in the experimental group, online word clouds and quizzes will be sent. All activities will be conducted at an appropriate time for the students.
  Interventions: Other: Flipped Learning
- Control group (No Intervention): Students who meet the inclusion criteria for the study will be administered the "Introductory Characteristics Form," the "Thoracic and Cardiac Examination Information Evaluation Form," and the "Self-directed Learning Skills Scale (SRLSS)" (pretest).
  Control group, the topic will be delivered using only traditional teaching methods. No additional resources will be provided to the students for preparation.
  The topic will be presented using a PowerPoint presentation, and question-answer sessions, demonstrations, and discussions will be conducted.
  After the presentation, and again 4 weeks later, the "Thorax and Heart Examination Knowledge Assessment Form" and the "Self-directed Learning Skills Scale (SRLSS)" will be administered to the both groups for evaluation (posttest).

INTERVENTIONS:
Other: Flipped Learning — Materials for students' pre-class studies and for use by the instructor during class will be created by the researchers. For students in the experimental group to come prepared for class according to the flipped learning model, digital materials will be prepared by the researchers. The experimental group will receive digital materials prior to the topic. The links to these materials will be sent to the students, who can access them via their mobile phones and watch the explanatory and demonstration videos as many times as they wish. Subsequently, the topic will be presented to the students. They will summarize the information learned from the videos and engage in question-answer sessions and discussions using prepared digital resources to address any points they do not understand. To reinforce the practices in the experimental group, online word clouds and quizzes will be sent.
  Arms: Flipped learning

SUMMARY:
This study is planned to determine the impact of education provided with the flipped learning model on nursing students' thorax and heart knowledge and self-directed learning skills. This study adopted a pretest-posttest openlabel randomized controlled trial. The population of the study will consist of second-year students studying at a Nursing Department of a university in Turkey during the 2023-2024 academic year.According to the power analysis, it was determined that the study needs to be conducted with a total of 100 students, with 50 students in the experimental group and 50 students in the control group.The experimental group participants were trained using the flipped learning model.For the control group, the topic will be delivered using only traditional teaching methods.The data for the study will be collected using the "Introductory Characteristics Form," the "Thoracic and Cardiac Examination Information Evaluation Form," and the "Self-Regulated Learning Skills Scale (SRLSS)."The collected data will be analyzed using SPSS 15 software.

DETAILED DESCRIPTION:
This study is planned to determine the impact of education provided with the flipped learning model on nursing students' thorax and heart knowledge and self-directed learning skills. Department of a Health Sciences Faculty. The population of the study will consist of second-year students studying at a Nursing Department of a university in Turkey during the 2023-2024 academic year. Power analysis was conducted to calculate the sample size of the study. G-Power 3.1.9.7 statistical software was used for the calculation of the sample size. The power analysis was based on a 5% error margin, 0.57 effect size, and 80% power level (Cohen, 1992). According to the power analysis, it was determined that the study needs to be conducted with a total of 100 students, with 50 students in the experimental group and 50 students in the control group.

Students who meet the inclusion criteria for the study will be administered the "Introductory Characteristics Form," the "Thoracic and Cardiac Examination Information Evaluation Form," and the "Self-directed Learning Skills Scale (SRLSS)" (pretest). Materials for students' pre-class studies and for use by the instructor during class will be created by the researchers.

For students in the experimental group to come prepared for class according to the flipped learning model, digital materials (such as lecture and demonstration videos) will be prepared by the researchers.

The experimental group will receive digital materials (such as explanatory and demonstration videos, Edpuzzle, etc.) prior to the topic. The links to these materials will be sent to the students, who can access them via their mobile phones and watch the explanatory and demonstration videos as many times as they wish.

Subsequently, the topic "Thorax and Heart Examination" will be presented to the students. They will summarize the information learned from the videos and engage in question-answer sessions and discussions using prepared digital resources to address any points they do not understand. To reinforce the practices in the experimental group, online word clouds and quizzes will be sent. All activities will be conducted at an appropriate time for the students.

For the control group, the topic will be delivered using only traditional teaching methods. No additional resources will be provided to the students for preparation. The topic will be presented using a PowerPoint presentation, and question-answer sessions, demonstrations, and discussions will be conducted.

After the implementation, and again 4 weeks later, the "Thorax and Heart Examination Knowledge Assessment Form" and the "Self-directed Learning Skills Scale (SRLSS)" will be administered to both the control and experimental groups for evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Second-year nursing students,
* Volunteer to participate in the research,
* Have continuous Internet Access
* Have smartphones/computers

Exclusion Criteria:

* Have previously studied in a health-related
* Have previously taken the physical examination course

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-16 (Estimated); Primary Completion 2025-01-17 (Actual); Study Completion 2025-01-17 (Estimated)

PRIMARY OUTCOMES:
The Thoracic and Cardiac Examination Information Evaluation Form | just before education, just after education, just 1 month after education
  This form, created based on the literature (Tuzer et al., 2016), includes pretest and posttest to measure the levels of knowledge about thoracic-lung and cardiac examinations. There are a total of 20 questions worth 100 points each related to thoracic and cardiac examinations in the tests. The questions in the tests consist of 20 multiple-choice questions.

SECONDARY OUTCOMES:
Self-Directed Learning Skills Scale | just before education, just after education, just 1 month after education
  The Self-Directed Learning Skills Scale (SDLSS) was developed by Tekkol and Demirel (2018). The scale consists of 21 items rated on a five-point Likert-type scale (always, usually, sometimes, rarely, and never). The scale has four subscales: self-monitoring, motivation, self-control, and self-confidence. Higher scores indicate higher self-directed learning skills. The scale has a Cronbach's alpha of 0.89 (Tekkol and Demirel, 2018), which was 0.85 (pretest), 0.89 (posttest), and 0.89 (follow-up testing) in the present study.

CONTACTS AND LOCATIONS:
Locations (1):
- Hilal Tuzer, Keçiören, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No